CLINICAL TRIAL: NCT03197441
Title: Intraoperative Platelet Rich Plasma Injection in Arthroscopic Surgery for Osteoarthritis of the Knee
Brief Title: Platelet Rich Plasma for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Superintendent, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-16028-RD-105065
Record Dates: First submitted 2017-04-13; First posted 2017-06-23 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Osteo Arthritis Knee; Platelet-rich Plasma
Keywords: Platelet-rich plasma; Osteoarthritis Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP group (Experimental): Arthroscopic knee surgery plus intraoperative platelet-rich plasma
  Interventions: Other: Platelet-rich plasma

INTERVENTIONS:
Other: Platelet-rich plasma — Intraoperative platelet-rich plasma injection during arthroscopic knee surgery

SUMMARY:
This study aimed to analyze the effect of platelet-rich plasma (PRP) on knee osteoarthritis. Eligible patients will undertake arthroscopic knee surgery plus intraoperative PRP and also receive second look surgery and intraoperative biopsy.

DETAILED DESCRIPTION:
Osteoarthritis is a chronic disease defined by progressive degradation of the joint as well as loss of cartilage on joint surfaces. The degeneration that occurs in the joint leads to changes in the catabolic and anabolic activity of chondrocytes. Osteoarthritis may induce pain, stiffness and limitation in range of motion of the joint and also may impact the quality of life. Platelet-rich plasma (PRP) is a fraction of plasma that contains platelets and multiple growth factors concentrated at high level. Because activated platelets have the potential to release growth factors, PRP has been clinically used to accelerate wound healing and tissue regeneration in orthopedic and oral surgery. Although several studies have assessed the effects of PRP on knee osteoarthritis, a higher level of evidence has not been provided. This study aimed to analyze the effect of PRP on knee osteoarthritis. After performing arthroscopic knee surgery plus intraoperative PRP in eligible patients, a second look arthroscopic surgery with intraoperative biopsy will be arranged 6 months later. Pre- and post-operative imaging and clinical outcomes will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 70 years
* With diagnosis of osteoarthritis, grade II~grade IV, II-III medial compartment

Exclusion Criteria:

* Lateral compartment and patellofemoral joint osteoarthritis
* With prior history of knee surgery
* Severe varus deformity
* With current or prior history of traum or infection at the knee
* With current or prior history of cancer
* With current or prior history of hematological disease
* Pregnancy
* Patients who will not cooperate with one-year followup

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Change in knee function from baseline to postoperative 3 months | 3-month postoperative
  Knee function is evaluated using Oswestry Disability Index preoperatively and 3-month postoperatively.

SECONDARY OUTCOMES:
Change in knee function from baseline to postoperative 6 months | 6-month postoperative
  Knee function is evaluated using Oswestry Disability Index preoperatively and 6-month postoperatively.
Change in knee function from baseline to postoperative 12 months | 12-month postoperative
  Knee function is evaluated using Oswestry Disability Index preoperatively and 12-month postoperatively.
Change in knee pain from baseline to postoperative 3 months | 3-month postoperative
  Pain is evaluated using visual analogue scale preoperatively and 3-month postoperatively.
Change in knee pain from baseline to postoperative 6 months | 6-month postoperative
  Pain is evaluated using visual analogue scale preoperatively and 6-month postoperatively.
Change in knee pain from baseline to postoperative 12 months | 12-month postoperative
  Pain is evaluated using visual analogue scale preoperatively and 12-month postoperatively.
Percentage of patients with regenerated cartilage | 12-month postoperative
  Cartilage regeneration is assessed by pathological biopsy during second look surgery at 12-month postoperative.
Change in cartilage thickness from baseline to postoperative 6 months | 6-month postoperative
  Cartilage thickness is assessed by MRI preoperatively and 6-month postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No